CLINICAL TRIAL: NCT06712173
Title: A Single Arm, Open Label, Single-center Dose-exploratory Clinical Study of Linperlisib in Combination With EZH2 Inhibitor SHR2554 in the Treatment of Relapsed/Refractory Peripheral T-cell Lymphoma
Brief Title: Linperlisib Combined With EZH2 Inhibitor in Relapsed/Refractory Peripheral T-cell Lymphoma (PTCL)
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2024029
Record Dates: First submitted 2024-11-25; First posted 2024-12-02 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Peripheral T Cell Lymphoma
Keywords: Peripheral T Cell Lymphoma; SHR2554; PI3K inhibitor linperlisib
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- linperlisib combined with SHR2554 (Experimental)
  Interventions: Drug: linperlisib and SHR2554

INTERVENTIONS:
Drug: linperlisib and SHR2554 — Linperlisib doses were preset at 40mg QD and 60mg QD, while SHR2554 doses were preset at 150mg BID, 200mg BID, and 300mg BID, forming six dose groups in total.

SUMMARY:
This is a Phase I, multicenter, non-randomized, open-label, dose-exploratory clinical study to evaluate the safety and tolerability of linperlisib combined with SHR2554 in the treatment of R/R PTCL, and to preliminary observe the antitumor efficacy of the combination of the two drugs.

DETAILED DESCRIPTION:
Linperlisib doses were preset at 40mg QD and 60mg QD, while SHR2554 doses were preset at 150mg BID, 200mg BID, and 300mg BID, forming six dose groups in total. The BOIN Waterfall design was employed to divide these six groups into two sub-trials.

Initially, three participants will be recruited into the lowest dose group of the first sub-trial: Linperlisib (40mg QD) and SHR2554 (150mg BID). After completing the dose-limiting toxicity (DLT) observation period, the next dose group will begin. Once DLT evaluations for the three participants are completed, the statistician will review the safety data and, following the decision-making flowchart of the BOIN design, determine whether to escalate to the next dose level. Another three participants will be enrolled and evaluated, continuing this process until all dose combinations in the first sub-trial have been tested, the sample size is depleted, or a stopping rule is triggered. Based on the results of the first sub-trial, the statistician will assess and select the starting dose for the second sub-trial, repeating the process until the trial is complete.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old, male or female;
2. Pathologically confirmed PTCL, including systemic anaplastic large cell lymphoma (ALCL), peripheral T cell lymphoma non-specific type (PTCL NOS), lymph node T-follicular helper cell lymphoma (nTFHL) [including nTFHL angioimmunoblastic type (NTFHL-AI), nTFHL follicular type (NTFHL-F) and nTFHL non-specific name (NTFHL-NOS)], enteropathy-associated T-cell lymphoma and hepato-splenic T-cell lymphoma;
3. Have received at least one previous systemic therapy, ALCL patients must have received CD30-targeted therapy; Patients were allowed to have received hematopoietic stem cell transplantation;
4. There must be at least one evaluable lesion/measurable lesion that meets the 2014 version of Lugano lymphoma evaluation criteria [Evaluable lesion
5. ECOG PS 0-2;
6. Adequate organ function:
7. Expected survival of at least 3 months;
8. Fertile male and female subjects are willing to use effective contraceptive measures throughout the study period and for six months after the last dose.
9. Volunteer to participate in clinical studies and sign informed consent, willing to follow and able to complete all trial procedures.

Exclusion Criteria:

If a patient has any of the following conditions should not be included in this study:

1. Had been treated with PI3K inhibitor or EZH2 inhibitor or EZH1/2 inhibitor before enrollment;
2. Primary cutaneous T-cell lymphoma;
3. History of other primary aggressive malignancies that are not in remission or in remission for no more than 3 years;
4. Involvement of the central nervous system (meninges or brain parenchyma);
5. People with a known allergy to any of the drugs in the study
6. Participated in other drug clinical trials within 4 weeks before the study began;
7. Pregnant or lactating women;
8. Active infected persons, except tumor-related B symptom fever;
9. Diseases and medical history:

   1. have multiple factors that affect oral medication (such as inability to swallow, chronic diarrhea and intestinal obstruction);
   2. have a history of psychotropic substance abuse and can not quit or have mental disorders;
   3. Subjects with any severe and/or uncontrolled medical condition;
10. A history of immunodeficiency, including HIV testing positive, or other acquired or congenital immunodeficiency diseases, or a history of organ transplantation;
11. Other situations deemed unsuitable for inclusion in the study by the researcher.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of linperlisib in combination with SHR2554 | 28 days since the date of first dose
  MTD will be established according to the incidence of dose-limiting toxicities (DLTs)

SECONDARY OUTCOMES:
Safety of linperlisib in combination with SHR2554 | From the start of treatment until 30 days after the last treatment
  The incidence and severity of treatment-emergent AEs will be collected and the safety and tolerability of linperlisib in combination with SHR2554 will be assessed.
Overall response rate (ORR) | 2 years
  Assess the response rate of subjects to the treatment of linperlisib in combination with SHR2554
Complete response (CR) rate | 2 years
  Assess the complete response rate of subjects to the treatment of linperlisib in combination with SHR2554
Progression-free survival (PFS) | 2 years
  Assess the survival condition of the subjects after the treatment of linperlisib in combination with SHR2554
Overall survival (OS) | 2 years
  Assess the overall survival of subjects treated by linperlisib in combination with SHR2554